CLINICAL TRIAL: NCT00936767
Title: Artemisone for the Treatment of Uncomplicated Falciparum Malaria in Western
Brief Title: Artemisone for the Treatment of Uncomplicated Falciparum Malaria in Western Cambodia
Acronym: AMOS
Status: Withdrawn | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Did not get approval
Sponsor: University of Oxford (Other)
Collaborators: Mahidol University (Other); Medicines for Malaria Venture (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BAKMAL0901
Record Dates: First submitted 2009-07-09; First posted 2009-07-10 (Estimated); Last update posted 2018-08-31 (Actual); Status verified 2010-10

CONDITIONS: Uncomplicated Falciparum Malaria
Keywords: falciparum malaria; artemisone; artesunate; resistance
MeSH Terms: conditions — Malaria, Falciparum | interventions — artemisone; Mefloquine; Artesunate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Artemisone/Mefloquine (AmiM3) (Experimental): Artemisone 4 mg/kg/day for 3 days plus mefloquine 15mg/kg on day 3 and 10mg/kg on day 4
  Interventions: Drug: Artemisone/Mefloquine (AmiM3)
- Artesunate/Mefloquine (MAS3) (Active Comparator): Artesunate 4mg/kg/day for 3 days plus mefloquine 15mg/kg on day 3 and 10mg/kg on day 4
  Interventions: Drug: Artesunate

INTERVENTIONS:
Drug: Artemisone/Mefloquine (AmiM3) — Artemisone 4 mg/kg/day for 3 days plus mefloquine 15mg/kg on day 3 and 10mg/kg on day 4
  Arms: Artemisone/Mefloquine (AmiM3)
Drug: Artesunate — Artesunate 4mg/kg/day for 3 days plus mefloquine 15mg/kg on day 3 and 10mg/kg on day 4
  Arms: Artesunate/Mefloquine (MAS3)

SUMMARY:
It has now been demonstrated clearly that in Western Cambodia parasitological responses to artesunate and artemether containing treatment regimens for uncomplicated falciparum malaria are slower than elsewhere in the world. Median parasite clearance time (PCT) in patients treated with artesunate 4 mg/kg/day was 78 hours and with 2 mg/kg/day 82 hours, compared to 54 and 48 hours, respectively, in Western Thailand; at 72hours peripheral blood parasitaemia was still detectable in 55% of patients in Western Cambodia, compared to 7.5% in Western Thailand. Although occasional poor responses to artesunate have been described previously the current reports suggest a consistent problem. These antimalarials are central to current treatment strategies, and so spread of parasites with reduced artemisinin susceptibility outside this area would be a disaster. A recent consensus meeting Pnomh Penh agreed that this should indeed be termed resistance, and represented a major threat to malaria control. Radical containment measures would be needed. This study aims to address whether a semi-synthetic or fully synthetic peroxide antimalarial would be more effective than artesunate and could therefore be used in Cambodia as part of the elimination strategy. Artemisone is a semisynthetic derivative of dihydroartemisinin, which importantly changes its tertiary structure. This drug has also shown promising efficacy for the treatment of uncomplicated falciparum malaria in phase II trials in Thailand and seems to be at least as efficacious as artesunate. No significant toxicity has been reported for artemisone and it is very well tolerated. If sensitivity for artemisone has remained intact in Western Cambodia, this will have important implications for the strategies available for containment of the threatening problem of artesunate resistance in Western Cambodia. It will also have important implications for further development of these drugs for the use in artemisinin combination therapies (ACTs).

DETAILED DESCRIPTION:
This is a small detailed randomised open-label clinical trial comparing the efficacy of oral artemisone with oral artesunate in the treatment of uncomplicated falciparum malaria in Western Cambodia. A detailed pharmacokinetic-pharmacodynamic evaluation and in vitro sensitivity for the study drugs will be part of the assessments. The overall design and proposed conduct is very similar to the recently completed studies of high dose artesunate.Fever patients in the villages surrounding Pailin (or equivalent study site) in Western Cambodia will be screened with a PfHRP2-based malaria rapid test (Paracheck) by the village malaria workers. In case of a positive test result, the patient will be transported by the study team to the hospital, full consent (as described above) and enrolment procedures will be conducted. It will be made clear from the outset that refusal to participate will in no way jeopardize subsequent antimalarial treatment.Eligibility can only be confirmed by a medically qualified investigator. Subjects who fulfil all the inclusion criteria and have none of the exclusion criteria will be randomised to one of the three treatment arms according to the randomisation schedule. Subject numbers will be will be assigned when the subject is enrolled after screening and prior to randomisation.Patients will be randomized in blocks of 15 to receive either artemisone 4 mg/kg/day for 3 days plus mefloquine 15mg/kg on day 3 and 10mg/kg on day 4 (N=50) or artesunate 4mg/kg/day for 3 days plus mefloquine 15mg/kg on day 3 and 10mg/kg on day 4 (N=25.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 16 years
* Full written informed consent is obtained
* Willingness and ability to comply with the study protocol for the duration of the trial including agreement to 5 days hospitalisation.
* History of fever or presence of fever (tympanic or axillary temperature at >37.5 °C).
* Peripheral blood P.falciparum parasitaemia between 10,000/uL and 200,000/uL. (Mixed malaria infection included)

Exclusion Criteria:

* Known hypersensitivity to the study drugs.
* Any antimalarial drug treatment in the 48 hours prior to enrolment.
* Clinical and/or laboratory features of severe malaria (as defined by WHO).
* Gastrointestinal dysfunction that could alter absorption or motility (i.e. active peptic ulcer, inflammatory bowel disease, malabsorption syndromes, intestinal sub-occlusion or previous major gastrointestinal surgery).
* Presence of intercurrent illness or any condition which in the judgement of the investigator would place the subject at undue risk or interfere with the results of the study.
* Splenectomy.
* Pregnant or lactating women. Serum test for β-HCG to be performed on any woman of child bearing age unless menstruating.
* Taking any contraindicated medicines (as listed in the most up to date product information)
* Participation in a clinical study within the previous 12 weeks
* Any other condition in the opinion of the investigator makes the patient unsuitable to be a subject

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-10; Primary Completion 2010-10 (Estimated); Study Completion 2010-10 (Estimated)

PRIMARY OUTCOMES:
Presence of light microscopic assessed peripheral blood parasitaemia at 72 hours after start of antimalarial treatment. | 72 hours

SECONDARY OUTCOMES:
Parasite clearance times (PCT, slope of the log clearance curve, PRR24, PRR48, PC50, PC90) | Variable
Cure rate defined as clearance of asexual parasites without recrudescence within a 28 and 63-day period. | 63 days
Number of adverse events | 9 weeks
Fever clearance time | Variable
In-vitro sensitivity to antimalarial drugs of P. falciparum from study patients | Day 0
Molecular determinants of antimalarial drug resistance. | Day 0
Pharmacokinetic parameters | Day 2
Hematocrit levels | Day 63
Gametocyte clearance | Variable

CONTACTS AND LOCATIONS:
Overall Officials: Duong Socheat, MD, Principal Investigator — Cambodia National Malaria Control Programme
Locations (1):
- Pailin Hospital, Pailin, Cambodia